CLINICAL TRIAL: NCT01101425
Title: Clinical and Biological Characterization of Male Breast Cancer: an International EORTC, BIG, TBCRC and NABCG Intergroup Study.
Brief Title: Male Breast Cancer: Understanding the Biology for Improved Patient Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Breast International Group (Other); Swiss Cancer Institute (Other); Cancer Trials Ireland (Network); Borstkanker Onderzoek Groep (Network); Swedish Association of Breast Oncologists (Unknown); Hellenic Cooperative Oncology Group (Other); Hellenic Oncology Research Group (Other); Latin American Cooperative Oncology Group (Other); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: EORTC-10085; BIG 2-07; TBCRC 029
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: male; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: Gathering medical information and tumor samples from patients with male breast cancer may help doctors learn more about the disease.

Purpose retrospective part: to perform a large international retrospective analysis of clinical and biological data of male BC patients treated in the participating centers from 1990 to 2010.

Purpose prospective part: to create a registry of men with breast cancer for a period of 30 months (starting early 2014).

DETAILED DESCRIPTION:
Objectives retrospective part (closed to patients registration in September 2013):

* To perform a large international joint retrospective analysis of clinical and biological data of male breast cancer (BC) patients treated from 1990 to 2010.
* To create a database of patient characteristics, disease features, treatments received, and clinical outcomes of a large series of men diagnosed with BC from 1990 to 2010 in centers in Europe and USA.
* To perform a central pathological review of the corresponding large series of male BC tumors to determine their biologic characteristics and identify relevant prognostic and predictive markers.

Objectives prospective part (opened early 2014):

* To run a prospective registry of all male BC patients (including newly diagnosed) irrespective of the stage and treatment, in the participating institutions for a period of 30 months; collection of FFPE, fresh frozen and blood samples is optional but highly encouraged.
* Quality of Life sub-study

The two parts of this study will provide important information regarding male BC biology and clinical evolution. The collected follow-up information will provide an overview of the current practice in the early and the advanced disease and also offer precious information of the disease evolution in such rare patients' population.

ELIGIBILITY:
Retrospective part (closed to patients registration):

* Men with histologically proven invasive breast carcinoma diagnosed since 1990 to 2010.
* A FFPE tissue sample from the primary tumor (e.g. biopsy or surgery) is mandatory

Prospective part:

* All men, with histologically proven invasive breast cancer, newly presenting at the center irrespective of the stage of disease, initial diagnosis date or treatment received.

  * patients cannot be registered in both the retrospective and protective parts of the study
  * patients who newly present at the center in the 3 months prior to center activation are still eligible as long as they were not previously included in the retrospective part of the study
* Before patient registration, written informed consent must be obtained according to ICH/GCP, and national/local regulations.
* Collection of left-over FFPE and frozen tumor samples as well as blood is optional.

Both parts:

* Concomitant DCIS or LCIS are allowed only if invasive cancer is present.
* Patients should be 18 years or over at the time of diagnosis.
* The study will accept all stages of disease (e.g. early BC, locally advanced and metastatic disease) independent of the treatment received. Patients with past or concurrent other malignancies are eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective part: males with histologically proven invasive breast carcinoma diagnosed since 1990 to 2010.
  Prospective part: all men, with histologically proven invasive breast cancer, newly presenting at the center irrespective of the stage of disease, initial diagnosis date or treatment received.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-12; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes: survival, progression free survival, time to locoregional relapse, time to distant relapse, time to second primary. | end of study
Patient and disease characteristics. | end of study
Patterns of treatment offered to these patients | end of study
Biological characterization of the disease | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Cardoso, MD, Study Chair — Champalimaud Cancer Center (Portugal); Sharon H. Giordano, MD, MPH, Study Chair — M. D. Anderson Cancer Center (TX, USA)
Locations (93):
- United States (17):
  - University Of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University Of Alabama Comprehensive Cancer Cente, Birmingham, Alabama
  - UCSF University of California San Francisco Medical Center-Mount Zion, San Francisco, California
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins University CRB1, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center - Memorial hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Baylor college of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Baylor College - Ucop, Houston, Texas
  - Fred Hutchison Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (12):
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU St Pierre, Brussels
  - Cliniques Universitaires St. Luc, Brussels
  - Hopital Universitaire Brugmann, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Hopital De Jolimont, Haine-Saint-Paul
  - UZ Leuven, Leuven
  - ZNA Jan Palfijn, Merksem
  - CHU Ucl Namu - Clinique Sainte Elisabeth, Namur
  - AZ Damiaan - Campus Sint-Jozef, Ostend
- Brazil (2):
  - Centro Regional Integrado de Oncologia, Fortaleza
  - Centro de Pesquisas Clinicas em Oncologia, Porto Alegre
- Ain Shams University Hospital, Cairo, Egypt
- Greece (10):
  - Alexandra Hospital, Athens
  - Aretaieio Hospital, Athens
  - General Hospital of Air Force, Athens
  - Hippokration General Hospital Of Athens, Athens
  - Hygeia Hospital, Athens
  - IASO general hospital, Athens
  - University General Hospital Heraklion, Heraklion
  - Agioi Anargiroi Hospital, Kifissia
  - General University Hospital Papageorgiou, Thessaloniki
  - Thermi Clinic, Thessaloniki
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordia Hospital, Dublin
  - St. James'S Hospital, Dublin
  - St. Vincent'S Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- Instituto Nacional De Cancerologia, México, Mexico
- BOOG, Amsterdam, Netherlands
- Instituto De Enfermedades Neoplasicas, Lima, Peru
- Poland (2):
  - Medical University Of Gdansk, Gdansk
  - Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw
- Portugal (2):
  - Champalimaud Cancer Center, Lisbon
  - Instituto Portugues De Oncologia - Centro Do Porto, Porto
- Institute of Oncology and Radiology, Belgrade, Serbia
- Spain (2):
  - Hospital General Vall D'Hebron, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- Swedish Association of Breast Oncologists, Gothenburg, Sweden
- Switzerland (16):
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Inselspital, Bern
  - Sonnenhofklinik Engeriedspital, Bern
  - Spitalzentrum Biel, Biel
  - Kantonales Spital Herisau, Herisau
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Cantonal Hospital Liestal, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital St Gallen, Sankt Gallen
  - ZeTuP St.Gallen, Sankt Gallen
  - Hopital de Sion, Sion
  - Radio-Onkologie Berner Oberland AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (18):
  - Worthing Hospital, Worthing, West Sussex
  - City Hospital, Birmingham
  - Royal Sussex County Hospital, Brighton
  - LLandough Hospital, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Leighton Hospital, Crewe
  - Queen Margaret Hospital, Dunfermline
  - Eastbourne District General Hospital, Eastbourne
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - New Victoria Hospital, Glasgow
  - Crosshouse Hospital, Kilmarnock
  - Forth Valley Royal Hospital, Larbert
  - Royal Liverpool University Hospital, Liverpool
  - Royal Alexandra Hospital, Paisley
  - University Hospital of North Tees, Stockton-on-Tees
  - The Great Western Hospital, Swindon
  - Wishaw General Hospital, Wishaw